CLINICAL TRIAL: NCT05497921
Title: Controlled Crossover Study to Evaluate the Efficacy of the handLITE LED Device in Treating the Signs of Contact/Irritant Dermatitis of the Hand
Brief Title: Crossover Study to Evaluate the Efficacy of LED in Treating the Signs of Contact/Irritant Dermatitis of the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Baker (Industry)
Responsible Party: Sponsor-Investigator, Steven Baker, Clinical Trial Manager, Ismart
Organization: Ismart (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASIRC_Hlcd06_02
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Contact Dermatitis of Hand

STUDY DESIGN:
Intervention Model Description: Subjects will treat one hand while the contralateral hand acts as a control. At the end of 6 weeks the subject will be instructed to cease treatment of the test hand and commence treatment of the control hand for 6 weeks. Efficacy will be evaluated at 6 weeks after the beginning of the treatment and 12 weeks (end of crossover).
Masking Description: PI will not know which is the treatment or control hand.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Test (device arm) (Other): Crossover study. The subject treats 1 hand while the contralateral is the control arm. After 6 weeks the treatment/control hand are swopped.
  Interventions: Device: handLITE LED device

INTERVENTIONS:
Device: handLITE LED device — handLITETM is a home use wearable LED phototherapy device. The device consists of a flexible silicone glove that contains red and near infrared light emitting diodes (LEDs) and a controller. The LEDs generate the light. The glove is worn on the hand and is held in place by an adjustable Velcro strap.

SUMMARY:
This study is intended to be a cross over study. Subjects will treat one hand while the contralateral hand acts as a control. At the end of 6 weeks the subject will be instructed to cease treatment of the test hand and commence treatment of the control hand for 6 weeks. Efficacy will be evaluated at 6 weeks after the beginning of the treatment and 12 weeks (end of crossover).

DETAILED DESCRIPTION:
This is a single-center study intended to be a cross-over study. Subjects will treat one hand while the contralateral hand acts as a control. At the end of 6 weeks, the subject will be instructed to cease treatment of the test hand and commence treatment of the control hand for 6 weeks. Efficacy will be evaluated at 6 weeks after the beginning of the treatment and 12 weeks (end of crossover). There will be no wash-out period during the crossover as this is not a systemic drug that has a half-life, and we expect subjects to still be exposed to the contact irritants. A crossover trial was chosen since this makes more use of a smaller trial group and removes the need for a separate parallel control group, therefore reducing trial numbers and allowing all subjects to be given the active treatment.

Since contact dermatitis is a chronic condition affected by external factors the skin condition should persist long enough for the investigator to expose the subject to the experimental treatment and measure the response. Since the subjects will still be exposed to their contact irritants as part of their daily life there should be no reason to introduce a washout period and since each subject acts as their own control, any systemic spread should be compensated for.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 21 and 75 years
* Subject with mild to moderate no greater than 50 on the SCORAD Index or 40 on the Objective SCORAD index stable contralateral contact/irritant dermatitis of the hand.
* Subjects agree to treat only one hand at a time for 6 weeks, the other acting as a control.
* 4-week washout period has elapsed since subject received topical treatments for contact/irritant dermatitis and oral antibiotics.
* Subjects agree to use a non-mediated soap substitute supplied for their use during the study period (Syndet)
* Subjects agree to NOT use any emollients 24 hours prior to their assessment days.

Exclusion Criteria:

* Subjects <21 and >75years of age.
* Subject with a grading score of > than 50 on the SCORAD Index or >40 on the Objective SCORAD index)
* The subject has lichenized or urticated papules or plaques.
* Subject has exudative atopic dermatitis
* Subject has localized infection
* Subjects currently taking prescriptive corticosteroids and antibiotics (topical or systemic).
* Subjects who have received PUVA or UVB therapy or any immunosuppressive therapy I the last 8 weeks.
* Planned exposure to sun, UVA or UVB that may affect the treatment area during the study period.
* Subjects who suffer from systemic photosensitive disorder such as Lupus erythematosus, photosensitive eczema, or Albinism.
* Subjects currently taking (or a history of taking) medication known to induce photosensitivity.
* Subjects who are pregnant or planning pregnancy during the study, breastfeeding mothers.
* Subjects enrolled in another clinical trial during the same study period.
* Subjects who have participated in a clinical trial in the last 30 days.
* Subjects who have a planned hospital admission and/or surgical procedure for an illness or disease which existed before enrolment into the clinical trial and which may interfere with the course or outcome of the study.
* Subjects who have a planned vacation that would exclude them from attending follow up evaluations.
* Subject has medical or psychological condition(s) associated with a risk of poor protocol compliance (e.g., alcoholism or drug abuse).
* Subject is undergoing or is likely to undergo other treatments.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction in the signs and symptoms of contact/irritant dermatitis of the hand according to a Modified SCORAD system | at 6-weeks
  eduction in the signs and symptoms of contact/irritant dermatitis of the hand according to a Modified SCORAD system

SECONDARY OUTCOMES:
Subjective assessment of treatment response (POEM) | At 6 weeks
  Subjective assessment of treatment response (POEM)

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, Principal Investigator — ASIRC
Locations (1):
- Dr Glynis Ablon MD, FAAD, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No